CLINICAL TRIAL: NCT04357327
Title: Rapid Salivary Test to Detect SARS-CoV-2 (COVID-19): a Diagnostic Accuracy Study
Brief Title: Rapid Salivary Test to Detect SARS-CoV-2 (COVID-19)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Lorenzo Azzi, Assistant Professor, Università degli Studi dell'Insubria
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 68/2020
Record Dates: First submitted 2020-04-15; First posted 2020-04-22 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: COVID-19; SARS-CoV 2; Corona Virus Infection
Keywords: SARS-CoV-2; COVID-19; Saliva; nCoV-2019; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Consecutive recruitment of both patients with COVID-19 like symptoms (i.e., cough, fever, dyspnea) and patients with low risk phenotype
Who Masked: Outcomes Assessor
Masking Description: The rapid salivary test will provide results within 5-10 minutes, while the rRT-PCR performed on nasopharyngeal swab shows results only after 6 hours, thus the outcome assessor of the experimental test is blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptomatic patients (Experimental): Patients with symptoms associated with COVID-19, i.e., dyspnea, cough, fever, etc.
  Interventions: Diagnostic Test: rapid salivary test
- Asymptomatic subjects (Active Comparator): Asymptomatic patients with low risk phenotype, that means patients with a previous negative swab, no relatives affected by COVID-19 and with reduced social interaction within the last two weeks.
  Interventions: Diagnostic Test: rapid salivary test

INTERVENTIONS:
Diagnostic Test: rapid salivary test — a rapid salivary test to detect SARS-CoV-2 spike protein in saliva with a lateral flow immunoassay

SUMMARY:
The present Diagnostic Accuracy study aims at experimentally validating the use of a rapid salivary test to detect SARS-CoV-2 infection in both symptomatic and asymptomatic individuals as a preliminary approach to a mass screening program.

The study is based on a consecutive recruitment of both patients showing symptoms probably associated with COVID-19 (i.e., cough, dyspnea, fever) and asymptomatic patients with a low risk phenotype. The expected number of recruited individuals is 100.

The experimental test is a prototype of salivary test based on the Lateral Flow Immunoassay technique and is able to detect the presence of SARS-CoV-2 in saliva, especially the Spike protein (S). The comparison is represented by the nasopharyngeal swab, the gold standard of COVID-19 diagnosis.

Patients will undergo both salivary immunoassay and nasopharyngeal swab, thus the outcome assessors are blinded, since the results of the rRT-PCR analysis require at least 6 hours before being available.

The main outcomes are sensibility and specificity of the rapid salivary test, when compared with the gold standard (nasopharyngeal swab).

ELIGIBILITY:
Inclusion Criteria:

People who undergo nasopharyngeal swab to confirm or exclude SARS-CoV-2 infection

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Sensibility | Salivary test will be interpreted after 10 minutes; the nasopharyngeal swab after 6 hours; sensitivity recorded through study completion, an average of 2 months.
  TP/TP+FN (TP= True Positive; FN = False Negative)
Specificity | Salivary test will be interpreted after 10 minutes; the nasopharyngeal swab after 6 hours; specificity recorded through study completion, an average of 2 months.
  TN/TN+FP (TN= True Negative; FP= False Positive)

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Azzi, Principal Investigator — Università degli Studi dell'Insubria
Locations (1):
- ASST dei Sette Laghi, Varese, VA, Italy

IPD SHARING:
Plan to Share IPD: Yes
We could provide anamnestic, clinical and serological data of each participant at the end of the study, or at least at the end of the first phase.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available at the end of the study, once statistical analyses is conducted
Access Criteria: Contact Principal Investigator